CLINICAL TRIAL: NCT05516875
Title: Open-Label Extension Study of JM-010 in Parkinson's Disease Patients With Dyskinesia
Brief Title: Open-Label Extension Study of ASTORIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial is terminated based on business decision, not due to safety concerns or regulatory requirements.
Sponsor: Contera Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JM-010CS-OL; 2022-002818-16 (EudraCT Number)
Record Dates: First submitted 2022-08-08; First posted 2022-08-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dyskinesias
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose (Experimental): JM-010 fixed combination drug (Group A) will be administered orally.
  Interventions: Drug: JM-010
- Low dose (Experimental): JM-010 fixed combination drug (Group B) will be administered orally.
  Interventions: Drug: JM-010

INTERVENTIONS:
Drug: JM-010 — JM-010

SUMMARY:
This current open-label extension (OLE) study (JM-010CS-OL) will explore the safety and tolerability of long-term administration of JM-010 of patients who completed 12-week treatment of Phase 2 (JM-010CS03) study.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to read, understand, and provide written, dated informed consent.
2. Subjects will be deemed likely to comply with study protocol and communicate with study personnel about adverse events (AEs) and other clinically important information.
3. Completed study visits per protocol in a previous JM-010CS03 study.
4. Ambulatory or ambulatory-aided (e.g. walker or cane) ability while ON, such that the subject can complete study assessments;
5. Knowledgeable and reliable caregiver/study partner, if appropriate, to accompany the subject to perform study visits and assist in completion of study instruments, as needed and allowed;
6. The subject himself/herself wishes to continue taking JM-010, and the investigator deems continued administration to be necessary or appropriate.

Exclusion Criteria:

1. Discontinued study drug in a previous JM-010 Dyskinesia efficacy study due to intolerable or unacceptable AEs considered to be related to JM-010.
2. Has other psychiatric (not including hallucinations due to side effects of dopamine therapy), neurological or behavioral disorders that in the opinion of the investigator may interfere with the conduct or interpretation of the study, including dementia, or subject who is considered violent.
3. Has a significant risk for suicidal behavior in the opinion of the investigator during the course of their participation in the study or

   * At Screening Visit: the subject scores "yes" on items 4 or 5 in the Suicidal Ideation section of the C-SSRS with reference to a 6-month period prior to Screening Visit; or
   * At Screening Visit: the subject has had 1 or more suicidal attempts with reference to a 2 year period prior to Screening Visit; or
   * At Baseline Visit: the subject scores "yes" on items 4 or 5 in the Suicidal Ideation section of the C SSRS with reference to Screening Visit
4. Has current seizure disorders (other than febrile seizures in childhood) requiring treatment with anti convulsants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant ECG abnormalities (Safety and Tolerability) | Baseline to Week 48
  12-lead electrocardiogram (ECG) assessments: Q-Tc interval in msec
Incidence of clinically significant cardiovascular abnormalities (Safety and Tolerability) | Baseline to Week 48
  Blood pressure in mmHg
Incidence of suicidal ideation or suicidal behavior (Safety and Tolerability) | Baseline to Week 48
  Columbia Suicide Severity Rating Scale (C-SSRS): Score ranges is 0- 50, where a higher score means more severe suicial ideation or behavior

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline to Week 48
  1. To summarize the efficacy of JM-010 in change in clinical progression of PD from Baseline to Week 48 as measured by the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS UPDRS) Parts I, Ⅱ, and Ⅲ.
  2. To summarize the efficacy of JM-010 in change in dyskinesia from Baseline to Week 48 as measured by the MDS-UPDRS Part IV.
  The score range is 0-132, where a higher score means more severe motor impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Contera Clinical Development, Study Director — Contera Pharma
Locations (2):
- Contera Investigational site_IT, Roma, Italy
- Contera Investigational site_ES, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No